CLINICAL TRIAL: NCT07102836
Title: COMPARATIVE EFFECTS OF ZINC AND PROBIOTICS ON NEONATAL INDIRECT HYPERBILIRUBINEMIA UNDERGOING PHOTOTHERAPY
Brief Title: COMPARISON OF ZINC AND PROBIOTICS ON NEONATES WITH INDIRECT HYPERBILIRUBINEMIA UNDERGOING PHOTOTHERAPY
Acronym: ZIPP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Quaid-e-Azam Medical College (Other)
Responsible Party: Principal Investigator, Malik Muhammad Umair Fazal, Dr. Malik Muhammad Umair Fazal, Quaid-e-Azam Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QAMC-CT-01; 248/DME/QAMC Bahawalpur (Other: DEPARTMENT OF MEDICAL EDUCATION QAMC BAHAWALPUR)
Record Dates: First submitted 2025-07-30; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Indirect Hyperbilirubinemia; Neonatal
Keywords: Zinc; Probiotics; Jaundice; Phototherapy; Neonates; Randomized Controlled Trial; Bilirubin; Enterohepatic Circulation; Indirect Hyperbilirubinemia
MeSH Terms: conditions — Jaundice | interventions — Zinc Sulfate; Zinc; Probiotics

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to two groups. One group will receive Zinc and other will be receiving Probiotics. This will be done in continuation of Phototherapy to compare the effects of both drugs in reducing indirect hyperbilirubinemia.
Who Masked: Participant, Care Provider
Masking Description: Both participants and care provider will be blinded to intervention allocation. Preparation of both drugs will be made identical in appearance and packaging to ensure unbiased administration and assessment during phototherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zinc group (Experimental): Participants in this group will receive oral zinc following neonatal dosing guidelines.
  Interventions: Drug: Zinc sulfate
- Probiotics group (Experimental): Participants in this group will receive oral probiotics following neonatal dosing guidelines.
  Interventions: Drug: Probiotic lactobacillus rhamnosus GG

INTERVENTIONS:
Drug: Zinc sulfate — Oral zinc sulfate syrup in a dose providing 5mg elemental zinc daily as adjuvant to phototherapy.
  Other Names: ZnSO4; Zinc
  Arms: Zinc group
Drug: Probiotic lactobacillus rhamnosus GG — Oral Probiotic Lactobacillus rhamnosus GG drops daily as adjuvant to phototherapy.
  Other Names: LGG; L. rhamnosus GG; Probiotic
  Arms: Probiotics group

SUMMARY:
Study will evaluate effects of oral zinc and probiotics supplementation in neonates who have indirect hyperbilirubinemia and are receiving phototherapy. Aim is to compare efficacy of these two drugs in clearing bilirubin and reducing duration of phototherapy. Neonates will be randomly assigned to receive either drug alongside phototherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Term or Near term neonates 2. Age <7 days at enrollment 3. Bilirubin levels within phototherapy range according to NICE bilirubin threshold charts 4. No identifiable pathology 5. Tolerating oral feeds 6. Parental or Guardian written informed consent taken.

Exclusion Criteria:

* 1. Positive sepsis screen or clinical signs of infection 2. Direct hyperbilirubinemia 3. Gastrointestinal malformations 4. Oral intolerance 5. Requiring mechanical ventilation 6. Congenital anomalies 7. Parental or Guardian refusal to participate in study

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2025-08-07 (Estimated); Primary Completion 2026-02-07 (Estimated); Study Completion 2026-05-07 (Estimated)

PRIMARY OUTCOMES:
Rate of decline in Bilirubin levels during phototherapy with this adjuvant therapy | From initiation of supplementation with phototherapy to its completion (typically 3-7 days).
  Primary outcome measures the rate at which total serum bilirubin decreases in mg/dL per day in neonates undergoing phototherapy while receiving supplementation with either zinc or probiotics. Bilirubin levels will be recorded at baseline and at regular intervals until phototherapy is discontinued and hence rate of decline will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Malik M. Umair Fazal, MBBS, FCPS Paediatrics, Principal Investigator — Quaid-e-Azam Medical College
Locations (1):
- Sadiq Abbasi Hospital, QAMC, Bahawalpur, Bahawalpur, Punjab Province, Pakistan